CLINICAL TRIAL: NCT03382925
Title: Do Cervical Interlaminar Epidural Steroid Injections With Low-dose Lidocaine Cause Transient Objective Upper Extremity Weakness? A Prospective Randomized
Brief Title: Does Low-does Cervical Epidural Lidocaine Cause Transient Weakness?
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Not enough cervical interlaminar patients who meet criteria in order to meet recruitment goals.
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Zack McCormick, Zachary L. McCormick, MD, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 106288
Record Dates: First submitted 2017-12-04; First posted 2017-12-26 (Actual); Results first posted 2021-05-18 (Actual); Last update posted 2022-11-25 (Actual); Status verified 2022-11

CONDITIONS: Cervical Radiculopathy
Keywords: cervical epidural steroid injection; local anesthetic; upper extremity weakness
MeSH Terms: conditions — Radiculopathy; Paresis | interventions — Lidocaine; Saline Solution; Triamcinolone Acetonide; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Masking Description: Each subject will be randomized into a group assignment in a 1:1 manner, #1 or #2, as outlined in the Methods section.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- cervical interlaminar with lidocaine (Active Comparator): Group #1: Interlaminar cervical ESI at the C7-T1 level with triamcinolone acetonide 80 mg (40 mg/mL) + 2 mL 1% lidocaine (total volume 4 mL).
  Interventions: Procedure: cervical interlaminar with lidocaine; Drug: Lidocaine; Drug: Triamcinolone Acetonide
- cervical interlaminar with normal saline (Active Comparator): Group #2: Interlaminar cervical ESI at the C7-T1 level with triamcinolone acetonide 80 mg (40 mg/mL) + 2 mL preservative saline (total volume 4 mL).
  Interventions: Procedure: cervical interlaminar with normal saline; Drug: Triamcinolone Acetonide; Drug: Normal saline

INTERVENTIONS:
Procedure: cervical interlaminar with lidocaine — Interlaminar cervical epidural steroid injection at the C7-T1 level with triamcinolone 80 mg (40 mg/mL) + 2 mL 1% lidocaine.
  Other Names: cervical epidural steroid injection
  Arms: cervical interlaminar with lidocaine
Procedure: cervical interlaminar with normal saline — Interlaminar cervical epidural steroid injection at the C7-T1 level with triamcinolone 80 mg (40 mg/mL) + 2 mL preservative saline
  Other Names: cervical epidural steroid injection
  Arms: cervical interlaminar with normal saline
Drug: Lidocaine — 2 mL lidocaine to be used as steroid diluent in group #1 cervical interlaminar procedure.
  Other Names: Xylocaine
  Arms: cervical interlaminar with lidocaine
Drug: Triamcinolone Acetonide — 2 mL of 40 mg/mL will be used as the steroid in group #1 and group #2 cervical interlaminar procedures.
  Other Names: Kenalog
Drug: Normal saline — 2 mL of normal saline to be used as steroid diluent in group #2 cervical interlaminar procedure.
  Other Names: sodium chloride
  Arms: cervical interlaminar with normal saline

SUMMARY:
"Does low-does cervical epidural lidocaine cause transient weakness?"

DETAILED DESCRIPTION:
Cervical radicular pain is relatively common, often treated with epidural steroid injection (ESI), when conservative treatments like oral analgesics, physical therapy, and activity modification have failed. There are no universal clinical practice guidelines for the use of diluents when CESI are performed.

Interlaminar CESI may be performed with or without the use of local anesthetics, due to training bias or theoretical concerns of weakness. CESI without the benefit of local anesthetic as a steroid diluent increases the latency of pain relief and may decrease diagnostic information immediately after a CESI with regard to pain generators responsible for symptoms, and may potentially decrease patient satisfaction.

By evaluating the effects of local anesthetic as a diluent during interlaminar cervical ESI, we will enhance the safety of this treatment with regard to expectations of objective motor weakness as well as post procedure pain control in the recovery phase after the injection procedure.

Additionally, investigation of short-term pain, function, medication use, and global impression of change following use of local anesthetic versus saline as a diluent during interlaminar cervical ESI will provide evidence to inform the optimization of clinical outcomes related to steroid diluent choice.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80.
2. Clinical diagnosis of cervical radicular pain.
3. Magnetic resonance imaging pathology consistent with clinical symptoms/signs.
4. Numerical Rating Scale (NRS) pain score of 4 or higher.
5. Pain duration of more than 6 weeks despite trial of conservative therapy (medications, physical therapy, or chiropractic care).
6. Patients who will undergo CESI for treatment of cervical radiculitis.

Exclusion Criteria:

1. Refusal to participate, provide consent, or provide communication and follow-up information for duration of the study.
2. Inability to perform handgrip or arm strength testing.
3. Contraindications to Cervical ESI (active infection, bleeding disorders, current anticoagulant or antiplatelet medication use, allergy to medications used for CIESI, and pregnancy).
4. Current glucocorticoid use or ESI within past 6 months.
5. Prior cervical spine surgery.
6. Cervical spinal cord lesions; cerebrovascular, demyelinating, or other neuro-muscular muscular disease.
7. Patient request for or requirement of conscious sedation for the injection procedure.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2019-08-19 (Actual); Study Completion 2020-08-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zachary L McCormick, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah Orthopaedic Center, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Peloso P, Gross A, Haines T, Trinh K, Goldsmith CH, Burnie S; Cervical Overview Group. Medicinal and injection therapies for mechanical neck disorders. Cochrane Database Syst Rev. 2007 Jul 18;(3):CD000319. doi: 10.1002/14651858.CD000319.pub4. PMID 17636629
- [Background] Stav A, Ovadia L, Sternberg A, Kaadan M, Weksler N. Cervical epidural steroid injection for cervicobrachialgia. Acta Anaesthesiol Scand. 1993 Aug;37(6):562-6. doi: 10.1111/j.1399-6576.1993.tb03765.x. PMID 8213020
- [Background] Ferrante FM, Wilson SP, Iacobo C, Orav EJ, Rocco AG, Lipson S. Clinical classification as a predictor of therapeutic outcome after cervical epidural steroid injection. Spine (Phila Pa 1976). 1993 May;18(6):730-6. doi: 10.1097/00007632-199305000-00010. PMID 8516703
- [Background] Botwin KP, Castellanos R, Rao S, Hanna AF, Torres-Ramos FM, Gruber RD, Bouchlas CG, Fuoco GS. Complications of fluoroscopically guided interlaminar cervical epidural injections. Arch Phys Med Rehabil. 2003 May;84(5):627-33. doi: 10.1016/s0003-9993(02)04862-1. PMID 12736872
- [Background] Rowlingson JC, Kirschenbaum LP. Epidural analgesic techniques in the management of cervical pain. Anesth Analg. 1986 Sep;65(9):938-42. PMID 3017152
- [Background] Castagnera L, Maurette P, Pointillart V, Vital JM, Erny P, Senegas J. Long-term results of cervical epidural steroid injection with and without morphine in chronic cervical radicular pain. Pain. 1994 Aug;58(2):239-243. doi: 10.1016/0304-3959(94)90204-6. PMID 7816491
- [Background] Lee SH, Kim KT, Kim DH, Lee BJ, Son ES, Kwack YH. Clinical outcomes of cervical radiculopathy following epidural steroid injection: a prospective study with follow-up for more than 2 years. Spine (Phila Pa 1976). 2012 May 20;37(12):1041-7. doi: 10.1097/BRS.0b013e31823b4d1f. PMID 22024908
- [Background] McCormick ZL, Nelson A, Bhave M, Zhukalin M, Kendall M, McCarthy RJ, Khan D, Nagpal G, Walega DR. A Prospective Randomized Comparative Trial of Targeted Steroid Injection Via Epidural Catheter Versus Standard C7-T1 Interlaminar Approach for the Treatment of Unilateral Cervical Radicular Pain. Reg Anesth Pain Med. 2017 Jan-Feb;42(1):82-89. doi: 10.1097/AAP.0000000000000521. PMID 27922950
- [Background] Capdevila X, Biboulet P, Rubenovitch J, Serre-Cousine O, Peray P, Deschodt J, d'Athis F. The effects of cervical epidural anesthesia with bupivacaine on pulmonary function in conscious patients. Anesth Analg. 1998 May;86(5):1033-8. doi: 10.1097/00000539-199805000-00024. PMID 9585292
- [Background] Bansal S, Turtle MJ. Inadvertent subdural spread complicating cervical epidural steroid injection with local anaesthetic agent. Anaesth Intensive Care. 2003 Oct;31(5):570-2. doi: 10.1177/0310057X0303100512. PMID 14601282
- [Background] Collier CB. Accidental subdural block: four more cases and a radiographic review. Anaesth Intensive Care. 1992 May;20(2):215-25. doi: 10.1177/0310057X9202000218. No abstract available. PMID 1317680
- [Background] Plastaras C, McCormick ZL, Garvan C, Macron D, Joshi A, Chimes G, Smeal W, Rittenberg J, Kennedy DJ. Adverse events associated with fluoroscopically guided lumbosacral transforaminal epidural steroid injections. Spine J. 2015 Oct 1;15(10):2157-65. doi: 10.1016/j.spinee.2015.05.034. Epub 2015 Jun 9. PMID 26065819
- [Background] Ortiz MP, Godoy MC, Schlosser RS, Ortiz RP, Godoy JP, Santiago ES, Rigo FK, Beck V, Duarte T, Duarte MM, Menezes MS. Effect of endovenous lidocaine on analgesia and serum cytokines: double-blinded and randomized trial. J Clin Anesth. 2016 Dec;35:70-77. doi: 10.1016/j.jclinane.2016.07.021. Epub 2016 Aug 6. PMID 27871598
- [Background] Gray A, Marrero-Berrios I, Weinberg J, Manchikalapati D, SchianodiCola J, Schloss RS, Yarmush J. The effect of local anesthetic on pro-inflammatory macrophage modulation by mesenchymal stromal cells. Int Immunopharmacol. 2016 Apr;33:48-54. doi: 10.1016/j.intimp.2016.01.019. Epub 2016 Feb 6. PMID 26854576
- [Background] van der Wal SE, van den Heuvel SA, Radema SA, van Berkum BF, Vaneker M, Steegers MA, Scheffer GJ, Vissers KC. The in vitro mechanisms and in vivo efficacy of intravenous lidocaine on the neuroinflammatory response in acute and chronic pain. Eur J Pain. 2016 May;20(5):655-74. doi: 10.1002/ejp.794. Epub 2015 Dec 18. PMID 26684648
- [Background] Bohannon RW. Reference values for extremity muscle strength obtained by hand-held dynamometry from adults aged 20 to 79 years. Arch Phys Med Rehabil. 1997 Jan;78(1):26-32. doi: 10.1016/s0003-9993(97)90005-8. PMID 9014953
- [Background] Bohannon RW. Grip strength impairments among older adults receiving physical therapy in a home-care setting. Percept Mot Skills. 2010 Dec;111(3):761-4. doi: 10.2466/03.10.15.PMS.111.6.761-764. PMID 21319615
- [Background] Hayes K, Walton JR, Szomor ZL, Murrell GA. Reliability of 3 methods for assessing shoulder strength. J Shoulder Elbow Surg. 2002 Jan-Feb;11(1):33-9. doi: 10.1067/mse.2002.119852. PMID 11845146
- [Background] Kolber MJ, Beekhuizen K, Cheng MS, Fiebert IM. The reliability of hand-held dynamometry in measuring isometric strength of the shoulder internal and external rotator musculature using a stabilization device. Physiother Theory Pract. 2007 Mar-Apr;23(2):119-24. doi: 10.1080/09593980701213032. PMID 17530541
- [Background] Awatani T, Mori S, Shinohara J, Koshiba H, Nariai M, Tatsumi Y, Nagata A, Morikita I. Same-session and between-day intra-rater reliability of hand-held dynamometer measurements of isometric shoulder extensor strength. J Phys Ther Sci. 2016 Mar;28(3):936-9. doi: 10.1589/jpts.28.936. Epub 2016 Mar 31. PMID 27134388
- [Background] Fieseler G, Molitor T, Irlenbusch L, Delank KS, Laudner KG, Hermassi S, Schwesig R. Intrarater reliability of goniometry and hand-held dynamometry for shoulder and elbow examinations in female team handball athletes and asymptomatic volunteers. Arch Orthop Trauma Surg. 2015 Dec;135(12):1719-26. doi: 10.1007/s00402-015-2331-6. Epub 2015 Sep 19. PMID 26386839
- [Background] Kirshblum SC, Waring W, Biering-Sorensen F, Burns SP, Johansen M, Schmidt-Read M, Donovan W, Graves D, Jha A, Jones L, Mulcahey MJ, Krassioukov A. Reference for the 2011 revision of the International Standards for Neurological Classification of Spinal Cord Injury. J Spinal Cord Med. 2011 Nov;34(6):547-54. doi: 10.1179/107902611X13186000420242. PMID 22330109
- [Background] Kim JK, Park MG, Shin SJ. What is the minimum clinically important difference in grip strength? Clin Orthop Relat Res. 2014 Aug;472(8):2536-41. doi: 10.1007/s11999-014-3666-y. Epub 2014 May 10. PMID 24817380

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cervical Interlaminar With Lidocaine | Cervical Interlaminar With Normal Saline
Started | 10 | 6
Completed | 10 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cervical Interlaminar With Lidocaine | Cervical Interlaminar With Normal Saline | Total
Number analyzed (Participants) | 10 | 6 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 6 | 14
  >=65 years | 2 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 5 | 2 | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 6 | 16

OUTCOME MEASURES:

1. Primary Outcome: Changes in Dynamometer Testing Post Procedure With Lidocaine vs Normal Saline.
Description: Strength Testing Dynamometry post procedure with lidocaine vs normal saline.
Time Frame: 30 minutes post-procedure
Population: Data was not collected. Study terminated early due to low enrollment. Zero participants completed both arms requirements. No statistical analysis obtained.
Arm/Group | Cervical Interlaminar With Lidocaine | Cervical Interlaminar With Normal Saline
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Sensory Exam Testing Post Procedure With Lidocaine vs Normal Saline.
Description: Sensory Exam of upper extremity
Time Frame: 30 minutes post-procedure
Population: as for outcome 1
Arm/Group | Cervical Interlaminar With Lidocaine | Cervical Interlaminar With Normal Saline
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Mean Arterial Blood Pressure Changes
Description: Mean Arterial Pressure
Time Frame: 30 minutes post-procedure
Population: as for outcome 1
Arm/Group | Cervical Interlaminar With Lidocaine | Cervical Interlaminar With Normal Saline
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Heart Rate Changes
Description: Heart Rate
Time Frame: 30 minutes post-procedure
Population: as for outcome 1
Arm/Group | Cervical Interlaminar With Lidocaine | Cervical Interlaminar With Normal Saline
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Pain Intensity
Description: Pain intensity will be measured by a 0-10 scale called Numerical Rating Scale. (0 being no pain and 10 being worst pain)
Time Frame: pre procedure, post-procedure, 1 day follow up, and one month follow up
Population: as for outcome 1
Arm/Group | Cervical Interlaminar With Lidocaine | Cervical Interlaminar With Normal Saline
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Upper Extremity Functional Index
Description: Upper Extremity Functional Index (UEFI) Questionnaire
Time Frame: pre procedure, post-procedure, 1 day follow up, and one month follow up
Population: as for outcome 1
Arm/Group | Cervical Interlaminar With Lidocaine | Cervical Interlaminar With Normal Saline
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Pain Medication
Description: Pain medication changes throughout treatment using MQS III calculator
Time Frame: pre procedure, post-procedure, 1 day follow up, and one month follow up
Population: as for outcome 1
Arm/Group | Cervical Interlaminar With Lidocaine | Cervical Interlaminar With Normal Saline
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Patient Global Impression of Change
Description: 7 point question called Patient Global Impression of Change
Time Frame: one month follow up
Population: as for outcome 1
Arm/Group | Cervical Interlaminar With Lidocaine | Cervical Interlaminar With Normal Saline
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected on each participant from their first day of enrollment until one month post procedure (Timeframe was approximately 1 1/2 months for each participant from enrollment, strength testing/procedure, to one month follow up). Duration of study enrollment was from December 20, 2017 to August 19, 2020 when study enrollment was closed.
Arm/Group | Cervical Interlaminar With Lidocaine | Cervical Interlaminar With Normal Saline
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/6
Serious Adverse Events (participants affected / at risk) | 1/10 | 0/6
Other Adverse Events (participants affected / at risk) | 0/10 | 0/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cervical Interlaminar With Lidocaine (N=10) | Cervical Interlaminar With Normal Saline (N=6)
Procedure AE (Cardiac disorders) | 1 (1) | 0 (0) — AE for cardiac and unrelated to procedure.

LIMITATIONS AND CAVEATS:
Early termination leading to low enrollment which ended up being the greatest limitation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-17): https://cdn.clinicaltrials.gov/large-docs/25/NCT03382925/Prot_SAP_000.pdf